CLINICAL TRIAL: NCT05861817
Title: Effect of Low Level Laser Therapy on Headache, and Fatigue in Patients With Chronic Rhinosinusitis.
Brief Title: Effect of Low Level Laser Therapy in Patients With Chronic Rhinosinusitis.
Acronym: Sinusitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Olfat Ibrahim Ali, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Chronic rhinosinusitis
Record Dates: First submitted 2022-05-28; First posted 2023-05-17 (Actual); Last update posted 2023-05-17 (Actual); Status verified 2023-05

CONDITIONS: Rhinosinusitis; Headache; Fatigue; CT
MeSH Terms: conditions — Rhinosinusitis; Headache; Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The participants were treated using LLLT (904nm and 2.5 J/ sinus) for one month
  Interventions: Device: Laser theapy
- Control group (Sham Comparator): using LLLT without output adjustment of the parameters
  Interventions: Device: Laser theapy

INTERVENTIONS:
Device: Laser theapy — participants were randomized into either the LLLT group or sham treatment group by a computer-generated random number. The participants were treated using LLLT (904nm and 2.5 J/ sinus). treatment was delivered for one month

SUMMARY:
This study aimed to evaluate the efficacy of low-level laser therapy (LLLT) for Chronic sinusitis in a randomized, double-blind, placebo-controlled trial.

DETAILED DESCRIPTION:
Chronic sinusitis, or chronic rhinosinusitis, is an inflammatory condition defined by symptomatic inflammation of the paranasal sinuses lasting longer than 3 months. Common presenting symptoms include nasal obstruction, facial pressure or fullness, nasal discharge (anterior or posterior), and olfactory loss. Furthermore, chronic sinusitis is associated with reductions in patient quality of life (QOL), sleep quality, and daily productivity.

It has been suggested that low-level laser can be used in treating chronic sinusitis but there are limited studies about its usage.

HYPOTHESES:

There is no statistically significant effect of laser therapy on headache, fatigue, or CT finding in patients with chronic sinusitis.

ELIGIBILITY:
Inclusion Criteria:

* patients suffering from mild to moderate symptoms.

Exclusion Criteria:

* Pregnant or breastfeeding women
* Patients with a definite deviated nasal septum, sinusitis, or history of operation within the last 6 months.
* Patients with hypertension, diabetes mellitus, malignancy, active pulmonary tuberculosis, infection, active respiratory disease like asthma, or other systemic diseases; • patients with long-term use of corticosteroids or immunosuppressive agents.
* Patients with hypersensitivity to the laser.
* Patients who were involved in another clinical study within 30 days.
* Patients who were unable to comply with the follow-up schedules.
* patients who had used antihistamines within 1 week, topical corticosteroids within2 weeks, systemic corticosteroids within 4 weeks, anti-cholinergic drugs within 3 days, antileukotriene drugs within 1 week, decongestants within 3 days, tricyclic antidepressants or phenothiazines within 2 weeks, non-steroidal analgesics within 2 weeks, and other drugs whi

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2022-01-18 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Headache | Baseline
  Headache was measured using headache scale at the beginning and end of the intervention. The scale ranged from zero to 10. The higher the scale the higher the headache
Headache | One month
  Headache was measured using headache scale at the beginning and end of the intervention. The scale ranged from zero to 10. The higher the scale the higher the headache

SECONDARY OUTCOMES:
Fatigue | Baseline
  Fatigue was measured using fatigue scale at the beginning and end of the intervention. The scale ranged from zero to 10. The higher the scale the higher the fatigue value.
Fatigue | One month
  Fatigue was measured using fatigue scale at the beginning and end of the intervention. The scale ranged from zero to 10. The higher the scale the higher the fatigue value.
Ct finding | Baseline
  number of sinus opacifications before and after intervention.
Ct finding | One month
  number of sinus opacifications before and after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Olfat I Ali, PhD, Principal Investigator — Cairo University
Locations (2):
- Egypt (2):
  - Faculty of physical therapy, Cairo university, Giza, Dokki
  - Olfat Ibrahim Ali, Giza, Dokki

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Abdulrashid NA, Ali OI, Elsharkawy MA. Effect of photobiomodulation therapy on headache, and fatigue in patients with chronic rhinosinusitis: a randomized controlled study. Lasers Med Sci. 2024 Feb 15;39(1):62. doi: 10.1007/s10103-024-04011-4. PMID 38358423